CLINICAL TRIAL: NCT05439928
Title: Remote Glucose Monitoring Using the Dexcom G6 Continuous Glucose Monitoring (CGM) System in Hospitalized Patients With Diabetic Ketoacidosis (DKA)
Brief Title: Remote Glucose Monitoring System in Hospitalized Patients With Diabetic Ketoacidosis (DKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Magdalena M. Bogun, MD, Assistant Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAT7802
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Ketoacidosis
Keywords: Continuous Glucose Monitoring; Diabetes; Hospitalized patients
MeSH Terms: conditions — Diabetic Ketoacidosis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DEXCOM G6 CGM (Experimental): Continuous glucose monitoring by DEXCOM G6 (glucose monitoring device) in a step-down unit in participants with DKA. This group comprises of both retrospective chart review and prospective patients.
  Interventions: Device: DEXCOM G6 CGM
- Hourly Finger Stick Point of Care (Historical Control) (No Intervention): DKA patients that received hourly glucose monitoring by finger stick while triaged through the ICU

INTERVENTIONS:
Device: DEXCOM G6 CGM — Continuous glucose monitoring
  Arms: DEXCOM G6 CGM

SUMMARY:
The purpose of this research study is to investigate the use of continuous glucose monitoring (CGM) device DEXCOM G6 in non-critically patients treated for diabetic emergency such as diabetic ketoacidosis (DKA). Patients who have DKA require hourly monitoring of glucose (sugar) level which traditionally requires admission to the intensive care unit (ICU) for hourly fingerstick monitoring. With the use of CGM device, in this research study hourly fingerstick monitoring is replaced by continuous glucose monitor (CGM) which provides glucose levels continuously in real time for nurses and provider. The investigators are testing to see if in the future patients can be treated in the stepdown unit (an intermediate care level between the intensive care unit and the general medical unit) if they do not require higher level of care besides hourly glucose monitoring. Continuous glucose monitoring (CGM) device DEXCOM G6 currently FDA Approved for patients with diabetes and is widely used for glucose monitoring in patients with diabetes in the outpatient setting. The investigators want to study the use of the DEXCOM G6 CGM in the inpatient setting to monitoring glucose levels remotely in the treatment of diabetic emergencies such as diabetic ketoacidosis and compare their care to those receiving hourly fingerstick glucose monitoring in the ICU.

DETAILED DESCRIPTION:
During the height of the COVID-19 pandemic, the investigators launched a quality improvement project with the goal of treating non-critically ill DKA patients outside of ICU setting to reallocate ICU beds for critically ill patients. The standard of care is for DKA patients to be treated in the ICU setting because the DKA protocol requires hourly fingerstick glucose monitoring, which is considered higher level of care and not appropriate for stepdown unit or medical/surgical wards. During this quality improvement project, the investigators monitored glucose levels remotely with continuous glucose monitoring (CGM) device DEXCOM G6, eliminating the need for hourly fingerstick glucose testing. Therefore, patients with DKA whose glucose levels were monitored with DEXCOM G6 CGM were treated in the stepdown unit instead of the ICU setting.

Once the number of COVID cases decreased and ICU beds were more readily available, the hospital returned to practicing pre-COVID standard of care, which was admitting DKA patient to the ICU for hourly glucose monitoring.

This study is a combined retrospective and prospective study of DKA patients. The investigators propose a retrospective chart review of DKA patients who had glucose levels monitored with DEXCOM G6 CGM during the COVID-19 pandemic. In the prospective portion of this study, participants will be enrolled and will undergo continuous glucose monitoring with DEXCOM G6 instead of the hourly fingerstick point of care glucose testing. Data collected for participants monitored via DEXCOM G6 (retrospective and prospective study data combined analysis) will be compared to participants with glucose levels monitored via hourly fingerstick in the ICU setting.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* AG>20 mEq/L
* Bicarbonate <15mEq/L
* Positive urine ketones or beta hydroxybutyrate >0.3 mmol/L

Exclusion Criteria:

* Hypotension (Blood Pressure below 80/60 mmHg)
* Requirement for pressor therapy
* Contraindication for utilizing Dexcom CGM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Bogun, MD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital/ Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group. Validation of measures of satisfaction with and impact of continuous and conventional glucose monitoring. Diabetes Technol Ther. 2010 Sep;12(9):679-84. doi: 10.1089/dia.2010.0015. PMID 20799388
- [Background] Nair BG, Dellinger EP, Flum DR, Rooke GA, Hirsch IB. A Pilot Study of the Feasibility and Accuracy of Inpatient Continuous Glucose Monitoring. Diabetes Care. 2020 Nov;43(11):e168-e169. doi: 10.2337/dc20-0670. Epub 2020 May 11. No abstract available. PMID 32393587
- [Background] Pasquel FJ, Umpierrez GE. Individualizing Inpatient Diabetes Management During the Coronavirus Disease 2019 Pandemic. J Diabetes Sci Technol. 2020 Jul;14(4):705-707. doi: 10.1177/1932296820923045. Epub 2020 May 5. PMID 32370606
- [Background] Chow KW, Kelly DJ, Rieff MC, Skala PA, Kravets I, Charitou MM, Morley EJ, Gupta R, Miller JD. Outcomes and Healthcare Provider Perceptions of Real-Time Continuous Glucose Monitoring (rtCGM) in Patients With Diabetes and COVID-19 Admitted to the ICU. J Diabetes Sci Technol. 2021 May;15(3):607-614. doi: 10.1177/1932296820985263. Epub 2021 Jan 12. PMID 33435706
- [Background] Davis GM, Galindo RJ, Migdal AL, Umpierrez GE. Diabetes Technology in the Inpatient Setting for Management of Hyperglycemia. Endocrinol Metab Clin North Am. 2020 Mar;49(1):79-93. doi: 10.1016/j.ecl.2019.11.002. PMID 31980123
- [Background] Umpierrez GE, Klonoff DC. Diabetes Technology Update: Use of Insulin Pumps and Continuous Glucose Monitoring in the Hospital. Diabetes Care. 2018 Aug;41(8):1579-1589. doi: 10.2337/dci18-0002. Epub 2018 Jun 23. PMID 29936424
- [Background] Newton CA, Smiley D, Bode BW, Kitabchi AE, Davidson PC, Jacobs S, Steed RD, Stentz F, Peng L, Mulligan P, Freire AX, Temponi A, Umpierrez GE. A comparison study of continuous insulin infusion protocols in the medical intensive care unit: computer-guided vs. standard column-based algorithms. J Hosp Med. 2010 Oct;5(8):432-7. doi: 10.1002/jhm.816. PMID 20945468
- [Background] Pal R, Banerjee M, Yadav U, Bhattacharjee S. Clinical profile and outcomes in COVID-19 patients with diabetic ketoacidosis: A systematic review of literature. Diabetes Metab Syndr. 2020 Nov-Dec;14(6):1563-1569. doi: 10.1016/j.dsx.2020.08.015. Epub 2020 Aug 18. PMID 32853901
- [Background] Li J, Wang X, Chen J, Zuo X, Zhang H, Deng A. COVID-19 infection may cause ketosis and ketoacidosis. Diabetes Obes Metab. 2020 Oct;22(10):1935-1941. doi: 10.1111/dom.14057. Epub 2020 May 18. PMID 32314455
- [Background] Fayfman M, Pasquel FJ, Umpierrez GE. Management of Hyperglycemic Crises: Diabetic Ketoacidosis and Hyperglycemic Hyperosmolar State. Med Clin North Am. 2017 May;101(3):587-606. doi: 10.1016/j.mcna.2016.12.011. PMID 28372715
- [Background] Livingston E, Desai A, Berkwits M. Sourcing Personal Protective Equipment During the COVID-19 Pandemic. JAMA. 2020 May 19;323(19):1912-1914. doi: 10.1001/jama.2020.5317. No abstract available. PMID 32221579

RESULTS

PARTICIPANT FLOW:
Groups:
- Hourly Finger Stick Point of Care (Historical Control): DKA patients that received hourly glucose monitoring by finger stick while triaged to the ICU.
Period: Overall Study
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control)
Started | 44 | 119
Completed | 44 | 119
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control) | Total
Number analyzed (Participants) | 44 | 119 | 163
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [33 to 66.5] | 47.66 [33.23 to 62.85] | 49.26 [33.23 to 63.34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 56 | 75
  Male | 25 | 63 | 88
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 44 | 119 | 163
Diabetes [Count of Participants; unit: Participants]
  Type 1 | 22 | 42 | 64
  Type 2 | 22 | 74 | 96

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Metabolic Acidosis
Description: Time to resolution of metabolic acidosis measured in hours. Resolution defined as anion gap (AG) <17 mEq/L and bicarbonate >19 mEq/L.
Time Frame: Up to 10 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control)
Number analyzed (Participants) | 44 | 119
hours | 12.84 [10 to 21.29] | 12.02 [8.33 to 22.68]

2. Secondary Outcome: Length of ICU Stay
Description: Length of ICU stay measured in days
Time Frame: Up to 20 days
Population: 60 participants in the Control group stayed in the ICU. No participants from the CGM group stayed in the ICU.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control)
Number analyzed (Participants) | 0 | 60
hours |  | 28.47 [20.86 to 48]

3. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay measured in hours
Time Frame: Up to 20 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control)
Number analyzed (Participants) | 44 | 119
hours | 120 [72 to 216] | 99.08 [72.73 to 150.73]

4. Secondary Outcome: Number of Hypoglycemic Events
Description: The number of hypoglycemic events will be recorded. A hypoglycemic event is defined as glucose level <70 mg/dL.
Time Frame: Up to 20 days
Measure: Number; unit: hypoglycemic events
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control)
Number analyzed (Participants) | 44 | 119
hypoglycemic events | 0 | 3

5. Other Pre Specified Outcome: Cost Savings
Description: Cost savings calculated by comparison of cost when non-critically DKA participants have glucose levels monitored via CGM and treated in the stepdown unit compared to participants who have glucose levels monitored via hourly fingersticks and treated in the ICU.
Time Frame: Up to 20 days
Population: Data was not collected
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 20 days
Arm/Group | DEXCOM G6 CGM | Hourly Finger Stick Point of Care (Historical Control)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/119
Other Adverse Events (participants affected / at risk) | 0/44 | 3/119
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEXCOM G6 CGM (N=44) | Hourly Finger Stick Point of Care (Historical Control) (N=119)
Hypoglycemic event defined as glucose level <70 mg/dL (Metabolism and nutrition disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT05439928/Prot_SAP_000.pdf